CLINICAL TRIAL: NCT06066437
Title: NeoAdjuvant Theranostic Lutetium Study: The Nautilus Trial
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Blue Earth Therapeutics (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0500; NCI-2023-08252 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-09-26; First posted 2023-10-04 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LeadIn: Treatment with 177Lu rhPSMA-10.1 (Experimental): Participants will receive 177Lu rhPSMA-10.1 alone.
  Interventions: Drug: Arm A: 177Lu rhPSMA-10.1; Drug: Arm B: 177Lu rhPSMA-10.1 plus Degarelix

INTERVENTIONS:
Drug: Arm A: 177Lu rhPSMA-10.1 — Participants will receive 177Lu rhPSMA-10.1 alone.
Drug: Arm B: 177Lu rhPSMA-10.1 plus Degarelix — Participants will receive 177Lu rhPSMA-10.1 alone. Participants will receive 177Lu rhPSMA-10.1 with Degarelix

SUMMARY:
To learn if the proposed dose of 177Lu rhPSMA-10.1 is safe. Phase 2 will open if the Phase 1 dose is found to be safe.

To learn about the safety and effects of 177Lu rhPSMA-10.1 alone and with androgen deprivation therapy (ADT) on patients with high-risk, localized prostate cancer before they have surgery to remove the disease.

DETAILED DESCRIPTION:
Primary Objectives:

The primary objective of the study is to assess safety and toxicity of 177Lu rhPSMA-10.1 Injection and to assess the impact of 177Lu rhPSMA-10.1 Injection with and without ADT on radiation dose delivered to the tumor in high risk localized and locoregional prostate cancer prior to primary radical prostatectomy with lymph node dissection.

Secondary Objectives:

* To assess the impact on pathologic outcomes at radical prostatectomy after 2 cycles of 177Lu rhPSMA-10.1 Injection with and without ADT Exploratory Objectives
* To evaluate the IHC expression of PSMA on pre-treatment prostate biopsy specimen compared to post ADT and 177Lu rhPSMA-10.1 Injectiontreatment surgical pathology
* To assess the impact on PSMA PET signal after treatment with 177Lu rhPSMA-10.1 Injection with and without ADT
* To evaluate efficacy of neoadjuvant 177Lu rhPSMA-10.1 Injection with or without ADT in men with high-risk and localized prostate cancer planned to undergo radical prostatectomy
* To evaluate exploratory predictive biomarkers for 177Lu rhPSMA-10.1 Injection with or without ADT including circulating tumor cells and extracellular vesicles

ELIGIBILITY:
Inclusion Criteria:

1. Men ≥18 years of age
2. Histologically documented prostatic adenocarcinoma with an NCCN risk group of high-risk or very high-risk. NCCN High Risk and Very High-Risk criteria shown below. (Network, N.C.C. (2021).

   Prostate Cancer (Version 02.2021).

   High Risk:
   * Has no very-high-risk features and has exactly one high-risk feature:
   * cT3a
   * Grade Group 4 or Grade Group 5
   * PSA >20 ng/mL

   Very high:
   * Has at least one of the following:
   * cT3b-cT4
   * Primary Gleason pattern 5
   * 2 or 3 high-risk features
   * >4 cores with Grade Group 4 or 5
3. Prostate biopsy within 90 days prior to randomization is allowed for entry requirements. Prostate biopsy must be reviewed at MD Anderson Cancer Center. Patients with small cell, neuroendocrine, or transitional cell carcinomas are not eligible
4. ECOG performance status (PS) grade 1
5. No evidence of metastatic disease or clinically positive lymph nodes as documented by technetium99m (99mTc) bone scan and by computed tomography (CT) or magnetic resonance imaging (MRI) scans. Imaging may be obtained up to 60 days prior to randomization
6. Minimum prostate tumor volume of 1.5 cm3 or greater as measured on prostate MRI within 60 days prior to randomization
7. Distant metastatic disease or clinically positive lymph nodes not identified by conventional imaging including by technetium-99m (99mTc) bone scan and by computed tomography (CT) or magnetic resonance imaging (MRI) scans but identified PSMA PET is allowed based on provider discretion
8. PSMA expression within the primary tumor with a minimum SUVmax of the primary tumor of at least 8
9. Localized or locally advanced disease deemed by the surgeon to be resectable. Patients must be appropriate candidates for and plan to undergo radical prostatectomy and pelvic lymph node dissection
10. No prior treatment for prostate cancer including prior surgery (excluding transurethral resection of the prostate [TURP]), cryoablation, pelvic lymph node dissection, radiation therapy, hormonal therapy or chemotherapy
11. Adequate bone marrow function documented by:

    * Hemoglobin ≥11 g/dL
    * Absolute neutrophil count ≥1.5 x 109/L
    * Platelet count ≥150 x 109/L
12. Adequate renal function defined as creatinine <1.5 x ULN or estimated glomerular filtration rate >60 mL/min/1.73 m2 using BSA with CKD-EPI
13. Adequate hepatic function documented by:

    * Total bilirubin ≤1.5 x ULN
    * AST ≤2.5 x ULN
    * ALT ≤2.5 x ULN
    * Alkaline Phosphatase (ALP) ≤2.5 x ULN

    Patients with Gilbert's syndrome do not need to meet total bilirubin requirements provided their total bilirubin is not greater than their historical level. Gilbert's syndrome must be documented appropriately as past medical history
14. Consents to providing whole blood samples for correlative PSMA evaluation of circulating tumor cells and extra cellular vesicles
15. Willing and able to comply with clinic visits and study-related procedures
16. Provide informed consent signed by study patient
17. To avoid risk of drug exposure through the ejaculate (even men with vasectomies), subjects must use a condom during sexual activity while on study drug and for 6 months following the last dose of study drug. If the subject is engaged in sexual activity with a woman of childbearing potential, a condom is required along with another effective contraceptive method consistent with local regulations regarding the use of birth control methods for subjects participating in clinical studies and their partners. Donation of sperm is not allowed while on study drug and for 3 months following the last dose of study drug.

Exclusion Criteria:

1. Prior hormone therapy for prostate cancer including orchiectomy, antiandrogens, ketoconazole, or estrogens (5-α reductase inhibitors allowed), or LHRH agonists/antagonists
2. Currently enrolled in another interventional study
3. Concurrent treatment with systemic corticosteroids (prednisone dose >10 mg per day or equivalent) or other immunosuppressive drugs <14 days prior to treatment initiation Steroids that are topical, inhaled, nasal (spray), or ophthalmic solution are permitted.
4. Known evidence of an active infection requiring systemic therapy such as uncontrolled human immunodeficiency virus (HIV), active hepatitis, or fungal infection. Uncomplicated urinary tract infection (UTI) does not qualify as an excluding infection.

   * Patients with HIV must be on an effective anti-retroviral regimen atleast four weeks prior to enrollment, HIV viral load less than 400 copies/mL and CD4+ T cell counts greater than 350 cell/uL.
   * Patients with HIV must agree to adhere to anti-retroviral therapy for the entirety of their participation in the protocol unless dictated by treatment toxicities.
   * Patients on Tenofovir will be excluded as there is a known risk of proximal renal tubule dysfunction leading to renal toxicity. Given that PSMA is expressed on the proximal tubule there is a theoretical risk of overlapping toxicity.
5. History of clinically significant cardiovascular disease including, but not limited to:

   * Myocardial infarction or unstable angina ≤6 months prior to treatment initiation
   * Clinically significant cardiac arrhythmia
   * Deep vein thrombosis, pulmonary embolism, stroke ≤6 months prior to treatment initiation
   * Congestive heart failure (New York Heart Association class III-IV)
   * Pericarditis/clinically significant pericardial effusion
   * Myocarditis
   * Endocarditis
6. History of major implant(s) or device(s), including but not limited to:

   * Prosthetic heart valve(s)
   * Current or prior history of infection or other clinically significant adverse event associated with an exogenous implant or device that cannot be removed
7. Other prior malignancy (exceptions: adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or any other cancer in situ currently in complete remission) ≤2 years prior to enrollment
8. Has received major surgery within 90 days of first administration of study drug
9. Prior allogeneic stem cell transplantation or recipients of organ transplants or autologous stem cell transplantation at any time MD Anderson Protocol Number: 2022-0500 2022-0500 Version Date 8/29/2023 26
10. Any medical, psychological or social condition that in the opinion of the investigator, would preclude participation in this study
11. Previously received external beam irradiation to the pelvis or to a field that includes more than 30% of the bone marrow or kidneys
12. Previous treatment with any of the following: PSMA-targeted radionuclide therapy, Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation
13. Transfusion of blood products for the sole purpose of meeting the eligibility criteria for this clinical trial
14. Patient has a functionally or anatomically solitary kidney.
15. Patients with Hydronephrosis and a Mag3 Lasix Renogram that demonstrates objective urinary obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average 1 year
Efficacy will be assess by measuring the radiation dose to the tumor (dosimetries) and PSA assessment | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chapin, M D, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org